CLINICAL TRIAL: NCT05279105
Title: Primary Health Care Landscape in Conflict Settings and Choices of Delivery Models in North West and South West Regions of Cameroon and North East Nigeria
Brief Title: Primary Health Care Delivery Models in Conflict Settings of Cameroon and Nigeria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Elrha (Other); Reach Out Cameroon (Unknown); University of Buea (Other); University of Maiduguri (Other); Herwa Community Development Initiative (HERWACDI) (Unknown)
Responsible Party: Principal Investigator, Lundi-Anne Omam Ngo Bibaa, PhD Candidate, University of Cambridge
Other Study IDs: Cambridge
Record Dates: First submitted 2022-02-17; First posted 2022-03-15 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Models of Care; Primary Health Care; Conflict-Affected Settings
MeSH Terms: interventions — Allied Health Personnel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Humanitarian workers: Staff working in humanitarian organisations will be recruited for interviews
  Interventions: Behavioral: Program support
- Internally displaced persons: Internally displaced persons living in conflict settings will be recruited for interviews
  Interventions: Behavioral: Program support

INTERVENTIONS:
Behavioral: Program support — The intervention to be evaluated in this study is program design and selection considerations by humanitarian organisations. It will comprise of factors that motivate organisations to chose certain delivery models in providing health care in conflict-affected settings

SUMMARY:
The overall objective of this research is to understand the PHC landscape in conflict-affected settings including choice of PHC delivery models and quality interventions used by humanitarian organisations

DETAILED DESCRIPTION:
There is sparse evidence to guide the selection and design of primary health care (PHC) services that improves and maintains quality care in humanitarian settings. The Northwest and Southwest regions of Cameroon, and Northeast Nigeria have protracted humanitarian crises. Various models of PHC are used in these settings; ensuring quality of PHC models of care is essential to improve health outcomes. We aim to explore how PHC models are selected by humanitarian organizations and through stakeholder engagement design a toolkit for evaluation of quality in PHC care delivery across different models.

The specific objectives of the study are;

1. To map different primary health care delivery models used by public, private and humanitarian organization in the conflict affected settings of NWSW Cameroon and North East Nigeria by conducting a mapping survey
2. To explore the factors influencing the selection of primary health care delivery models used by humanitarian organizations to guide the selection of models of care and strengthening of programming efforts in conflict settings by conducting an exploratory qualitative study
3. To determine the coverage and gaps in services across the different PHC models to develop a pilot questionnaire to evaluate quality in conflict settings by conducting an exploratory qualitative study

The humanitarian crisis in North West and South West regions of Cameroon and North East Nigeria, has led to the closure of 269/933 and 617/2367 health facilities respectively with over 2.21 million IDPs and 350,000 returnees(2, 3), creating a huge gap in the availability and accessibility of health services to affected communities. The need to conduct this study becomes even more pertinent to inform program developers and donors on key considerations to make before using different models of care, and how quality can be improved to foster sustainability

ELIGIBILITY:
Inclusion Criteria:

* Male and female staff of humanitarian organisations, internally displaced persons (confirmed to be a resident of an IDP or host community);
* Age 21 years of age or older;
* Ability to provide informed consent or assent to participate in the research

Exclusion Criteria:

* Individuals who are mentally ill or with limitations to communicate well;
* Those who cannot speak or understand the local languages so that they cannot understand the interviewer.
* Those who refuse to provide consent to the study or who do not want to participate in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Study population will be adults of age 21 years and above. The research will be undertaken with staff of humanitarian organizations and internally displaced populations. Project managers, project supervisors, grant writers and frontline workers of humanitarian organizations (UN agencies, international NGOs, national NGOs and CBOs) will be interviewed. Internally displaced persons in urban, peri-urban, rural and hard-to-reach areas. We will purposefully select participants from across the geographical area to ensure wide coverage of experiences/ views. In Cameroon and Nigeria, regions and states will be divided between rural, peri-urban and urban, and humanitarian organisations implementing programs in these areas will be group into urban, peri-urban and rural responders.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of frameworks developed | 12 months
  Framework to guide humanitarian organizations in the selection of primary health care models will be collaboratively developed following the results from the study and stakeholders meeting

SECONDARY OUTCOMES:
Number of quality oversight toolkit developed | 12 months
  Following the development of a framework to inform the selection of models of care, an "oversight toolkit" for selecting models of care and monitoring a pragmatic set of quality interventions (QI) will be developed. The toolkit will include a composite score drawing from scores across all domains. This will be used to give an overall assessment score of quality.

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Parkes-Ratanshi, Principal Investigator — University of Cambridge
Locations (3):
- Reach Out Cameroon, Buea, South-West Region, Cameroon
- Herwa Cdi, Maiduguri, Nigeria
- Lundi-Anne Omam Ngo Bibaa, Cambridge, United Kingdom